CLINICAL TRIAL: NCT02406794
Title: Effect of Kinesiotaping for the Treatment of Hormone-induced Myalgia in Women: Randomised Controlled Trial
Brief Title: Effect of Kinesiotaping for the Treatment of Hormone-induced Myalgia in Women Given Breast Cancer Survivors
Acronym: KITMYCAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Professor of Faculty of Health Sciences, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FCCSS-UMA_01-13
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2016-10

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Hormonal therapy; Aromatase inhibitors; Estrogen deprivation; Myalgia; Arthralgia; Carpal tunnel syndrome; Pressure pain threshold; Neuromuscular taping; Kinesio taping
MeSH Terms: conditions — Breast Neoplasms; Myalgia; Arthralgia; Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuromuscular taping (Experimental): The first group will receive a decalogue of healthy tips (general, to lead an active life) based on the best available evidence, and several strips of neuromuscular bandage will be applied on areas that refer pain (cervical, lumbosacral, both or wrist-forearm).
  Interventions: Drug: Neuromuscular taping
- No Kinesio taping (No Intervention): No Kinesio taping

INTERVENTIONS:
Drug: Neuromuscular taping — The first group will receive a decalogue of healthy tips (general, to lead an active life) based on the best available evidence, and several strips of neuromuscular bandage will be applied on areas that refer pain (cervical, lumbosacral, both or wrist-forearm).
  Other Names: Kinesio taping
  Arms: Neuromuscular taping

SUMMARY:
Background: It has been demonstrated that aromatase inhibitors (AIs) are more effective than tamoxifen in reducing breast cancer recurrence. However, despite the excellent results, the side effects associated with them cause between 24.5 and 31.3% therapy abandon. This study aimed to verify the effectiveness of Neuromuscular Taping (NMT) in the treatment of myalgia and arthralgia induced by AIs in women who have had breast cancer. Our goal is to improve their pain, decreasing by 20% the values of their Visual Analogue Scale (VAS) at various points in order to improve symptoms and increase adherence.

Methods/Design: The study includes 156 breast cancer survivors treated with endocrine therapy (aromatase inhibitors or tamoxifen and aromatase inhibitors) from Virgen de la Victoria Hospital (Málaga, Spain) and musculoskeletal disorders resulting from such treatment. Clinical and patient data were obtained from medical histories, genetic and proteomic analysis, grip strength and algometry measured, questionnaires and the outcome of interest, their VAS. NMT is applied in four possible locations, according to the symptoms of each participant: carpal tunnel, cervical, lumbar or lumbar and cervical. There are several more interventions before repeating the readings from the last five weeks of the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* To be of legal age
* Having suffered from primary breast cancer with histological confirmation (I-IIIA)
* Completion of primary carcinoma treatment (surgery, chemotherapy, radiotherapy)
* To be receiving hormone therapy as an adjunct to the process by aromatase inhibitors (exemestane, anastrozole, letrozole)
* To present a functional status according to WHO from 0 (asymptomatic, complete and ambulatory activity) or 1 (symptomatic but completely ambulatory, strenuous physical activity restricted but able to perform sedentary gentle activities)
* To understand correctly Spanish
* To show their approval by signing the informed consent
* Having had musculoskeletal disorders attributable to IA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Medical questionnaire | 10 minutes
  A record will be kept of some medical data such as tumor grade, types carried, complementary treatments and end date, and the type of hormone therapy received and start date. The possible presence of comorbidities will also be collected.
  Genetic determinants. Analyze genetic determinants due to the importance of genetic background on AIA and abandonment of therapy (Garcia-Giralt N., 2013). Estrogen receptor 1 (ESR1), aromatase (CYP19A1) and steroid, 17-alpha-hydroxylase / 17,20 lyase (CYP17A1) (Garcia-Giralt N., 2013), (Henry NL, 2012) and (Mao JJ, 2011) have been selected as candidate genes.
  Samples for extracting genes will be collected in both cases with controls on the baseline and the end of it. The DNA is extracted from whole blood using the DNA Blood Maxi Qiafilter (Qiagen, Inc., Valencia, CA) (Henry NL, 2013) kit.

SECONDARY OUTCOMES:
Sociodemographic and anthropometric questionnaire | 10 minutes
  This questionnaire will contain information on the following variables: gender and date of birth, marital status... Add basic anthropometric data such as weight, height, BMI, waist circumference and hip.
Plasma proteins (or proteomic analysis) | 10 minutes
  For our analysis investigators use four plasma proteins: serum amyloid A, collectin, immunoglobulin G (IgG) light chain kappa and add C1Q (Minton O., 2013).
PPT | 10 minutes
  The pain threshold pressure is defined as the minimum amount of pressure with which an initial feeling of pressure switches to pain. (Vanderweeën L. 1996). PPT measurements were performed on:
  * Cervical Musculature in space interapofisario C5-C6.
  * Lumbosacral Musculature: an L4 level on the erector spinae muscle.
  * Median nerve as it passes through the carpal bones.
Grip strength as measured by a Dynamometer | 5 minutes
  This instrument will be used to measure grip strength of both upper limbs. This test of strength has been previously used to measure the loss of strength in breast cancer survivors (Kaya T, 2010), even in cases where patients were treated with IAs (Lintermans A., 2011) . The dynamometer has proven to be the safest [ICC = 0.98] and most valid [ICC = 0.99] method to measure grip strength of the hand. (Bellace JV, 2000).
POMS | 10 minutes
  This is a scale to measure the profile of mood states. It consists of 65 items with five possible answers. The questionnaire delivered to patients is frequently used for study of breast cancer survivors (Cantarero-Villanueva, 2011). The reliability of the Spanish version of the POMS is high (Cronbach's α ranging from .76 to 0.91).
quality of life as assessed by QuickPIPER questionnaire | 10 minutes
  Tool used to determine the degree of perception that cancer patients have of their feelings of fatigue and how it alters their quality of life.
  This short version of the questionnaire proved to be adequate, with values of Kaiser-Meyer-Oklin (0.89) and Bartlett's sphericity test (P <0.001) index. The goodness of fit indices of confirmatory factor analysis are (normed fit index = 0.91 and = 0.92 comparative rate setting) satisfactory. The test-retest reliability of this questionnaire is very good (r = 0.947, P <0.001). (AI Cuesta-Vargas, 2013).
EORTC QLQ-C30 | 10 minutes
  This is a specific questionnaire for cancer, "core", created by the EORTC Group. It consists of 30 items to assess HRQOL and physical, emotional, social status and overall functioning of patients diagnosed with cancer. The questions refer to the last week from the date on which the respondent completed the form. It is organised in several multi-item scales and some independent items. The reliability of the QLQ-C30 is adequate, with Cronbach Alpha values between 0.52 and 0.89 in different scales. (Moro D.,2011)
pain as measured by VAS | 10 minutes
  The Visual Analogue Scale (VAS) was designed to allow a subjective assessment of pain. A VAS is usually a horizontal line of 10 cm. with perpendicular lines at the ends, which are defined as the extreme limits of the painful experience. Previous studies have shown that the VAS has adequate psychometric properties, including test-retest reliability (r = 0.78) and convergent validity with other measures of pain such as the McGill Pain Questionnaire (r = 0.49 to 0.65) (Sriwatanakul K ., 1983).
SFI-Sp | 10 minutes
  For this study we will use the Spanish version (SFI-Sp), since it has proven to be a valid and reliable measure of the spinal region result. This regional tool reflects the status and any change in the kinetic chain of the spine. This questionnaire has demonstrated high internal consistency (α = 0.85) and reliability (r = 0.96) (AI Cuesta-Vargas, 2014).
ULFI-Sp | 10 minutes
  This study uses the Spanish version (ULFI-Sp). This questionnaire has demonstrated high internal consistency (α = 0.94) and reliability (r = 0.93), making it a very useful tool for the evaluation of patients with disorders of the upper limbs, in both the clinical and research fields (AI Cuesta-Vargas, 2013).
BADIX | 10 minutes
  This Index includes a score for five movements of the trunk upright that result in Back Pain Index (BAI) and a record of "Morning Stiffness in the Back" (MBS). The sum of the BAI and MBS gives the BADIX (max. 20 points) (Kovacs FM, 2002).
  The BADIX appears to be a valid and reliable tool for the evaluation of morning stiffness restricting the mobility of the back, and discriminates whether the result of a treatment has been successful or not. (Farasyn A., 2013).
  This new Back Pain Disability index seems reliable (test-retest after 3 days) and is valid in the case of significant clinical change; it has also been shown to have discriminatory power and effect size comparable to other indices in assessing disability of patients with low back pain sensitivity. (Farasyn A., 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Study Director — University of Malaga; Inmaculada Conejo-Tirado, Principal Investigator — University of Malaga
Locations (1):
- Regional University Hospital Virgen de la Victoria, Málaga, Malaga, Spain

REFERENCES:
- [Derived] Conejo I, Pajares B, Alba E, Cuesta-Vargas AI. Effect of neuromuscular taping on musculoskeletal disorders secondary to the use of aromatase inhibitors in breast cancer survivors: a pragmatic randomised clinical trial. BMC Complement Altern Med. 2018 Jun 11;18(1):180. doi: 10.1186/s12906-018-2236-3. PMID 29890985